CLINICAL TRIAL: NCT01861717
Title: A Pilot Study of Pre- and Post-operative Somatuline Depot Therapy in Acromegalic Patients Treated by Endonasal Endoscopic Surgery: Impact on Early Remission Rates and Perioperative Morbidity
Brief Title: A Pilot Study of Pre- and Post-operative Use of Somatuline Depot.
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Didn't enroll enough subjects
Sponsor: Saint John's Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KELD-ESS-0413
Record Dates: First submitted 2013-05-15; First posted 2013-05-24 (Estimated); Results first posted 2021-09-30 (Actual); Last update posted 2021-09-30 (Actual); Status verified 2021-09

CONDITIONS: Acromegaly
Keywords: excess growth hormone; excess GH; gigantism; pituitary tumor; pituitary adenoma; growth hormone tumor; GH secreting adenoma; Somatuline; lanreotide
MeSH Terms: conditions — Acromegaly; Gigantism; Pituitary Neoplasms | interventions — lanreotide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Somatuline Depot Subcutaneous (SC) (Experimental): Somatuline Depot SC 90mg deep subcutaneous injection every 4 weeks for 3 doses before surgery. The dose will be 60 mg for patients with mild liver or kidney dysfunction.
  Interventions: Drug: lanreotide

INTERVENTIONS:
Drug: lanreotide — Somatuline Depot 90 mg deep subcutaneous injection every 4 weeks X 3 doses
  Other Names: Somatuline Depot SC

SUMMARY:
If someone is diagnosed with a pituitary tumor that causes acromegaly (too much growth hormone) the treatment is to have it surgically removed. This study has two phases.

The first phase provides medical treatment with a drug that will be provided for 3 months before surgery to see if complications of surgery are reduced and to see whether or not remission improves following surgery if you have this medical treatment. The drug administered is approved by the FDA for long-term treatment of acromegaly. It is not routinely administered before surgery, and is therefore experimental as used in this way. All other procedures performed during this research are standard of care with the exception of the 3 questionnaires to be completed at each visit.

The second phase of this study is from 3 months until 12 months after surgery and is only for people who do not go into remission after the operation. This phase assesses the possible remission of acromegaly after resuming the drug treatment for an additional 3 to 9 months. The drug will be prescribed by your physician as part of your regular medical care and will not be included as part of the study. All other procedures performed during this research are standard of care with the exception of the 3 questionnaires to be completed at each visit.

The study lasts approximately 16 months - 3 month before surgery and 12 months after surgery.

ELIGIBILITY:
Inclusion Criteria:

* age 18 - 75
* elevated serum Insulin-like growth factor-1 (IGF-1) level above age- and sex-based normal values and failure of growth hormone(GH) suppression to < 1.0 ng/ml after a 75 gm oral glucose tolerance test (OGTT) American Association of Clinical Endocrinolgists (AACE) Acromegaly Clinical Guidelines 2004
* visible pituitary adenoma (microadenoma or macroadenoma) on high quality pituitary MRI without and with gadolinium
* prior treatments for acromegaly with surgery, somatostatin analogs or pegvisomant are acceptable if these therapies have been discontinued for at least 3 months prior to study entry

Exclusion Criteria:

* Age < 18 or > 75 years
* acromegalic patients currently on a lanreotide or octreotide preparation or on pegvisomant
* patients who have received prior radiotherapy or radiosurgery
* patients with adenoma-related visual acuity or visual field deficit from optic nerve and/or chiasm compression or severe optic nerve/chiasm compression in the setting of normal visual fields and acuity
* patients with pituitary apoplexy defined as recent tumor hemorrhage and/or infarction on MRI with associated symptoms of new onset visual loss, diplopia and/or adrenal insufficiency

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2013-05 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniel F Kelly, MD, Principal Investigator — Saint John's Cancer Institute
Locations (1):
- Brain Tumor Center and Pituitary Disorders Program, John Wayne Cancer Institute, Saint John's Health System, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Brain Tumor Center and Pituitary Disorders Program, John Wayne Cancer Institute at Saint John's Health Center — http://newstjohns.org/braintumorcenter.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited between May 2013 and January 2016, in outpatient cancer center clinic
Groups:
- Somatuline Depot Subcutaneous (SC): Somatuline Depot Subcutaneous (SC) 90mg deep subcutaneous injection every 4 weeks for 3 doses before surgery. The dose will be 60 mg for patients with mild liver or kidney dysfunction.
  lanreotide: Somatuline Depot 90 mg deep subcutaneous injection every 4 weeks X 3 doses
Period: Overall Study
Arm/Group | Somatuline Depot Subcutaneous (SC)
Started (started = signed consent) | 4
Completed | 2
Not Completed | 2
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: Consented to participate in study
Groups:
- Somatuline Depot SC: Somatuline Depot SC 90mg deep subcutaneous injection every 4 weeks for 3 doses before surgery. The dose will be 60 mg for patients with mild liver or kidney dysfunction.
  lanreotide: Somatuline Depot 90 mg deep subcutaneous injection every 4 weeks X 3 doses
Arm/Group | Somatuline Depot SC
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: Early Remission of Acromegaly
Description: Early remission status after a 12 week course of pre-operative Somatuline Depot and 3 months after endonasal endoscopic surgery. Remission status will be based on age-adjusted Insulin Glucose Factor 1 (IGF-1) levels and oral glucose tolerance test.
Time Frame: 3 months post-op
Population: 2 patients treated; data not analyzed because study terminated prematurely.
Arm/Group | Somatuline Depot Subcutaneous (SC)
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Cardiac Function
Description: Changes in cardiac function after 12 weeks of Somatuline therapy and 3 months after endonasal endoscopic adenoma removal.
Time Frame: 3 month post-op
Population: 2 patients treated; data not analyzed because study terminated prematurely.
Arm/Group | Somatuline Depot SC
Number analyzed (Participants) | 0

3. Secondary Outcome: Change in Hypertension
Description: Change in hypertension after 12 weeks of Somatuline therapy and 3 months after endonasal endoscopic adenoma removal
Time Frame: 3 months
Population: 2 patients treated; data not analyzed because study terminated prematurely.
Arm/Group | Somatuline Depot SC
Number analyzed (Participants) | 0

4. Secondary Outcome: Change in Respiratory Function
Description: Change in respiratory function after 12 weeks of Somatuline therapy and 3 months after endonasal endoscopic adenoma removal
Time Frame: 12 weeks and 3 months
Population: 2 patients treated; data not analyzed because study terminated prematurely.
Arm/Group | Somatuline Depot SC
Number analyzed (Participants) | 0

5. Secondary Outcome: Change in Quality of Life
Description: Change in Quality of Life after 12 weeks of Somatuline therapy and 3 months after endonasal endoscopic adenoma removal
Time Frame: 3 months
Population: 2 patients treated; data not analyzed because study terminated prematurely.
Arm/Group | Somatuline Depot SC
Number analyzed (Participants) | 0

6. Other Pre Specified Outcome: Remission Status 1 Year After Surgery
Description: Remission status one year after surgery and time to achieve remission in patients who did not achieve remission after endonasal endoscopic surgery and who had resumption of Somatuline Depot therapy 3 months after surgery.
Time Frame: 12 months post-op
Population: 2 patients treated; data not analyzed because study terminated prematurely.
Arm/Group | Somatuline Depot SC
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 15 months
Arm/Group | Somatuline Depot SC
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Somatuline Depot SC (N=2)
Headache (Nervous system disorders) | 2 (2)
weight loss (Investigations) | 1 (1)
urinary frequency (Renal and urinary disorders) | 2 (2)
abdominal pain (Gastrointestinal disorders) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 1 (1)
blurred vision (Eye disorders) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 (1) — ears feel full of water
pain (General disorders) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) — due to blood loss during surgery
Dysgeusia (Nervous system disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 1 (1)
fatigue (General disorders) | 1 (1)
Nervous system disorders - Other, specify (Nervous system disorders) | 1 (1) — anosmia

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes